CLINICAL TRIAL: NCT02417779
Title: Effects of Extracorporeal Shock Wave Therapy in Cutaneous Microcirculation of Different Wounds
Brief Title: Cutaneous Microcirculation After Extracorporeal Shock Wave Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Kisch, MD, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-266-1
Record Dates: First submitted 2015-03-12; First posted 2015-04-16 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Burn Injury; Acute Wound; Chronic Wound; Burn Scar; Flap Disorder
MeSH Terms: conditions — Burns | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (12):
- Second-Degree Burn (Experimental): Group A (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Skin Excision (for Skin Graft) (Experimental): Group B (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size must not be less than 1% of TBSA.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Chronic Wound (Experimental): Group C (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Intact Skin (Active Comparator): Group D (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups A-C must be evident.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Second-Degree Burn (repetitive) (Experimental): Group E (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.
  Intervention: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Skin Excision (for Skin Graft) (repetitive) (Experimental): Group F (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size must not be less than 1% of TBSA.
  Intervention: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Chronic Wound (repetitive) (Experimental): Group G (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.
  Intervention: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Intact Skin (repetitive) (Active Comparator): Group H (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups A-C must be evident.
  Intervention: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Hypertrophic burn scar (Experimental): Group I (n=20): Consent-capable male and female patients ≥18 years of age suffering from a hypertrophic burn scar.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Hypertrophic burn scar (repetitive) (Experimental): Group J (n=20): Consent-capable male and female patients ≥18 years of age suffering from a hypertrophic burn scar.
  Intervention: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Flap (Experimental): Group K (n=20): Consent-capable male and female patients ≥18 years of age who received a flap.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Flap (repetitive) (Experimental): Group L (n=20): Consent-capable male and female patients ≥18 years of age who received a flap.
  Intervention: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave) — Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Arms: Chronic Wound; Flap; Hypertrophic burn scar; Intact Skin; Second-Degree Burn; Skin Excision (for Skin Graft)
Device: Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave) — Repetitive Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Arms: Chronic Wound (repetitive); Flap (repetitive); Hypertrophic burn scar (repetitive); Intact Skin (repetitive); Second-Degree Burn (repetitive); Skin Excision (for Skin Graft) (repetitive)

SUMMARY:
In plastic and reconstructive surgery, treatment strategies of second-degree burns, superficial wounds, hypertrophic burn scars, flaps and chronic wounds aim at reducing infection and improving microcirculation. Although previous studies indicate that extracorporeal shock wave therapy (ESWT) can accelerate wound healing, only a few studies focused on the elucidation of its mechanisms of action. Therefore, the aim of this study is to evaluate the microcirculatory effects of extracorporeal shock wave therapy on second-degree burns, superficial wounds, hypertrophic burn scars, flaps and chronic wounds in a human in-vivo setting for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Group A (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.
* Group B (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of TBSA.
* Group C (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.
* Group D (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups A-C must be evident. No soft tissue injury must be evident.
* Group E (n=20): Consent-capable male and female patients ≥18 years of age who have sustained a second-degree burn on ≥1% and ≤30% of the surface of the body.
* Group F (n=20): Consent-capable male and female patients ≥18 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of TBSA.
* Group G (n=20): Consent-capable male and female patients ≥18 years of age suffering from a wound that has not yet healed ≥3 weeks. The minimal size of the wound site must not be less than 1% of TBSA.
* Group H (n=20): Consent-capable healthy male and female probands ≥18 years of age serving as sham group. None of the the criteria of groups E-G must be evident. No soft tissue injury must be evident.
* Group I (n=20): Consent-capable male and female patients ≥18 years of age suffering from a hypertrophic burn scar.
* Group J (n=20): Consent-capable male and female patients ≥18 years of age suffering from a hypertrophic burn scar.
* Group K (n=20): Consent-capable male and female patients ≥18 years of age who received a flap.
* Group L (n=20): Consent-capable male and female patients ≥18 years of age who received a flap..

Exclusion Criteria:

General exclusion criteria

* below 18 years of age
* wounds requiring artificial respiration, since consent for the study participation is unobtainable

Exclusion Criteria Groups A, B, D, E, F, H:

* peripheral arterial occlusive disease
* vasculitis
* diabetes mellitus
* chronic kidney or liver disease
* cardiac dysfunction
* arterial hypo- or hypertension

Anamnestic exclusion criteria

* ongoing immunosuppressive or chemotherapy treatment
* drug abuse
* systemic skin diseases
* systemic and local cortisone therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Change in microcirculation (composite measure) | Baseline and 1 minute post-dose
  * capillary blood flow [arbitrary units AU]
  * capillary blood velocity [AU]
  * tissue oxygen saturation [%]
  * relative postcapillary venous filling pressure [AU]

SECONDARY OUTCOMES:
Change in microcirculation (areolar measure) | Baseline, while and 1 minute post-dose
  * tissue oxygen saturation [%]
  * tissue hemoglobin index

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany